CLINICAL TRIAL: NCT05716048
Title: Randomized Controlled Trial of Combined Cognitive Rehabilitation and Exercise Training for Learning and Memory in Persons With Moderate to Severe Traumatic Brain Injury
Brief Title: Combinatory Rehabilitation Used for Substantially Helping Individuals With Traumatic Brain Injury
Acronym: CRUSH-IT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Brian Sandroff, Senior Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-1195-22
Record Dates: First submitted 2023-01-13; First posted 2023-02-08 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KF-mSMT Plus Aerobic Exercise Training (Experimental): Participants will undergo 12 weeks of supervised aerobic cycling exercise training. During the last 8 weeks of cycling exercise, participants will also undergo treatment with the Kessler Foundation modified Story Memory Technique as an approach for cognitive rehabilitation.
  Interventions: Behavioral: KF-mSMT Plus Aerobic Exercise Training
- KF-mSMT Plus Stretching Exercise Training (Active Comparator): Participants will undergo 12 weeks of supervised stretching and toning exercise training. During the last 8 weeks of stretching exercise, participants will also undergo treatment with the Kessler Foundation modified Story Memory Technique as an approach for cognitive rehabilitation.
  Interventions: Behavioral: KF-mSMT Plus Stretching Exercise Training

INTERVENTIONS:
Behavioral: KF-mSMT Plus Aerobic Exercise Training — Participants will undergo this combinatory intervention 3 days per week for 12 weeks. The combined session duration will begin with 15 minutes and last up to 2 hours by the end of the 12th week
  Arms: KF-mSMT Plus Aerobic Exercise Training
Behavioral: KF-mSMT Plus Stretching Exercise Training — Participants will undergo this combinatory intervention 3 days per week for 12 weeks. The combined session duration will begin with 15 minutes and last up to 2 hours by the end of the 12th week
  Arms: KF-mSMT Plus Stretching Exercise Training

SUMMARY:
New learning and memory impairment (NLMI) is a common and devastating manifestation of TBI associated with substantial life burdens. Persons with moderate to severe TBI have shown improvement in NLM for prose material (e.g. story) as well as beneficial changes in default-mode network (DMN) activation during list-learning19 following treatment with the Kessler Foundation modified Story Memory Technique® (KF-mSMT®). Benefits, however, were moderate and did not yield downstream improvements in daily life. It is thus critical to examine other approaches to complement the KF-mSMT® for robustly managing NLMI in TBI. The proposed RCT will be the first to include aerobic exercise training (AET) as a highly-promising complement to the KF-mSMT® for robustly managing NLMI, examining impact on NLM, its neural correlates, and daily life in NLM impaired persons with moderate-to-severe TBI. We thus propose a two-arm, parallel group, double-blind RCT comparing the effects of the KF-mSMT+AET with the KF-mSMT+S/T (active control condition) on NLM (Aim 1), hippocampal MRI (Aim 2), and daily life outcomes (Aim 3). 60 NLM impaired persons with moderate-to-severe TBI will be randomized to one of 2 conditions (30 per condition). Each condition will take place 3 days per week for 12 weeks and will be supervised by KF personnel. Participants will be blinded as to the intent of the conditions. We will further explore baseline predictors of clinically meaningful changes in NLM for those completing the KF-mSMT + AET condition (Exploratory Aim 4). If successful, this trial will position combinatory KF-mSMT and AET within the clinician's arsenal for robustly managing NLMI in persons with TBI. By augmenting the effects of KF-mSMT with AET, this treatment aims to exert a powerful countermeasure to TBI-related NLMI, and ultimately help those with TBI-related NLMI return to the workforce, independently manage their everyday lives, and maintain optimal quality of life. Additionally, while rigorously designed to answer the scientific question of the relative benefit of AET with the KF-mSMT, the proposed study is will likely provide some level of benefit to all study participants.

If successful, this trial will provide Class I evidence of combined KF-mSMT and AET for rehabilitating NLMI in TBI, based on standards published for therapeutic trials by the American Academy of Neurology, thus positioning such an approach within the clinician's arsenal for robustly managing NLMI. By augmenting the effects of KF-mSMT with AET, we anticipate this treatment will ultimately help those with TBI-related NLMI return to the workforce, independently manage their everyday lives, and maintain optimal quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 to control for age related brain changes
* Diagnosis of moderate-to-severe TBI based on TBIMS criteria at least one year prior to enrollment
* Having no to low substance use / involvement (drug/alcohol) as documented via ASSIST
* Being insufficiently physically active based on a Godin Leisure-Time Exercise Questionnaire Health Contribution Score of <14
* Having a proficiency in the English language
* Being right handed to control for brain organization
* Having chronic medical conditions (e.g. diabetes) in addition to TBI will require approval to participate from a physician, consistent with PAR-Q+.
* Having an in-tact ability to follow directions based on the Telephone Interview for Cognitive Status (TICS-M) (i.e., TICS-M scores of ≥18)
* Demonstrating new learning and memory impairment based on Open-Trial Selective Reminding Task (OT-SRT) scores at least 1.5 standard deviations below healthy controls (8+ trials to reach criterion)

Exclusion Criteria:

* Regularly taking steroids & benzodiazapines to control for medications effects
* Having a history of neurological disorders beyond TBI
* Having a history of severe mental illness (e.g., schizophrenia, bipolar, severe major depression)
* Having metal in the body, claustrophobia, and other risk factors that would make MRI scanning unsafe.
* Having moderate or high risk for exercise training contraindications (e.g. diabetes), defined as ≥1 YES on pages 2-3 of the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+)
* Having significantly impaired vision by scotomas (corrected vision in worse eye worse than 20/60), diplopia, or nystagmus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in California Verbal Learning Test-3 Performance | From 0 to 12 weeks
  This is a test of new learning and memory

SECONDARY OUTCOMES:
Change in hippocampal volume | From 0 to 12 weeks
  This involves a structural MRI scan wherein the volume of the bilateral hippocampi will be measured.
Change in hippocampal activation | From 0 to 12 weeks
  This involves an fMRI list-learning task wherein activation of the hippocampus during encoding and recall will be measured
Change in hippocampal resting-state functional connectivity | From 0 to 12 weeks
  This involves a resting-state fMRI paradigm wherein connectivity between the hippocampus and other brain regions that are important for learning and memory will be measured.
Change in Everyday Memory Simulations Performance | From 0 to 12 weeks
  This multi-component test examines aspects of memory that are relevant to daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D Chiaravalloti, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided